CLINICAL TRIAL: NCT03140085
Title: Bacteriophages for Treating Urinary Tract Infections in Patients Undergoing Transurethral Resection of the Prostate: A Randomized, Placebo-controlled, Double-blind Clinical Trial
Brief Title: Bacteriophages for Treating Urinary Tract Infections in Patients Undergoing Transurethral Resection of the Prostate
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Principal Investigator, Thomas Kessler, Dr., Balgrist University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02/283
Record Dates: First submitted 2017-04-27; First posted 2017-05-04 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Intravesical Bacteriophage Treatment for Urinary Tract Infections
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anbiotica (Active Comparator)
  Interventions: Drug: Antibiotics
- Bacteriophages (Active Comparator)
  Interventions: Biological: PYO Phage
- Placebo (Placebo Comparator)
  Interventions: Other: Sterile bacteriology media

INTERVENTIONS:
Biological: PYO Phage — Intravescial instillation
  Arms: Bacteriophages
Drug: Antibiotics — Oral application
  Arms: Anbiotica
Other: Sterile bacteriology media — Sterile bacteriology media, with identical color as bacteriophage preparation
  Arms: Placebo

SUMMARY:
Urinary tract infections are among the most prevalent microbial diseases and their financial burden on society is substantial. The use of bacteriophages against bacterial pathogens has gained over the last years a renewed interest, because of the continuing increase in antibiotic resistance worldwide. Thus, the aim of this study is to investigate the efficacy of intravesical bacteriophage treatment to normalize urine culture compared to intravesical placebo or standard antibiotic treatment in a randomized controlled trial following a pilot phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urinary tract infections who are scheduled for transurethral resection of the prostate with urine culture (taken by mid-stream urine; or from the existing transurethral or suprapubic catheter) ≥104 colony forming units /mL of predefined uropathogens, including Enterococcus spp., Escherichia coli, Proteus mirabilis, Pseudomonas aeruginosa, Staphylococcus spp., and Streptococcus spp. and lower urinary tract symptoms such as urgency, frequency, dysuria, increased number of incontinence episodes
* Written informed consent.

Exclusion Criteria:

* Fever >38°C
* CRP >100mg/L
* Acute prostatitis
* Concomitant fungal urinary tract infection
* Current antibiotic treatment or antibiotic treatment within the last 7 days (exceptions: subjects with an active catheter associated urinary tract infection who have received prior antibiotics may be enrolled provided a minimum of 48 hours has elapsed between the last dose of the prior antibiotic and the time of obtaining the baseline urine specimen. Subjects receiving current antibiotic prophylaxis for catheter associated urinary tract infection who present signs and symptoms consistent with an active new catheter associated infection may be enrolled provided all other eligibility criteria are met including obtaining a pre-treatment qualifying baseline urine culture)
* Any rapidly progressing disease or immediately life-threatening illness including but not limited to: acute hepatic failure, respiratory failure, and septic shock
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Normalisation of urine culture | 7 days after treatment
  Success of intravesical treatment, defined as normalization of urine culture (no evidence of bacteria, i.e. <104 colony forming units/mL) after 7 days of bacteriophage, placebo, or antibiotic treatment

SECONDARY OUTCOMES:
Urine culture | Baseline and 7 days after treatment
Bladder diary | Baseline and 7 days after treatment
  Assessment of number of voids, number of leakages, post void residual
Pain diary | Baseline and 7 days after treatment
  Visual analog scale (0 (no pain) to 10 (strongest possible pain))
IPSS questionnaire | Baseline and 7 days after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- National Center of Urology, Tbilisi, Georgia

REFERENCES:
- [Derived] Leitner L, Ujmajuridze A, Chanishvili N, Goderdzishvili M, Chkonia I, Rigvava S, Chkhotua A, Changashvili G, McCallin S, Schneider MP, Liechti MD, Mehnert U, Bachmann LM, Sybesma W, Kessler TM. Intravesical bacteriophages for treating urinary tract infections in patients undergoing transurethral resection of the prostate: a randomised, placebo-controlled, double-blind clinical trial. Lancet Infect Dis. 2021 Mar;21(3):427-436. doi: 10.1016/S1473-3099(20)30330-3. Epub 2020 Sep 16. PMID 32949500
- [Derived] Leitner L, Sybesma W, Chanishvili N, Goderdzishvili M, Chkhotua A, Ujmajuridze A, Schneider MP, Sartori A, Mehnert U, Bachmann LM, Kessler TM. Bacteriophages for treating urinary tract infections in patients undergoing transurethral resection of the prostate: a randomized, placebo-controlled, double-blind clinical trial. BMC Urol. 2017 Sep 26;17(1):90. doi: 10.1186/s12894-017-0283-6. PMID 28950849